CLINICAL TRIAL: NCT05174858
Title: Efficacy of a Collagen Topical Hemostatic Agent After Tooth Extraction: a Comparative Randomized Clinical Trial
Brief Title: Efficacy of a Collagen Hemostatic Dressing After Tooth Extraction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ACTEON Group (Industry)
Collaborators: Slb Pharma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ETIKOL; 2021-A02568-33 (Other: French National Agency oh Health (ANSM))
Record Dates: First submitted 2021-12-13; First posted 2022-01-03 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Tooth Avulsion
Keywords: Hemostasis; tooth extraction; oral surgery; human
MeSH Terms: conditions — Tooth Avulsion

STUDY DESIGN:
Intervention Model Description: Study subject will be randomized in a 1:1 allocation ratio between the 2 treatment groups
Who Masked: Participant
Masking Description: the participant will be blind from the treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Device under investigation (Experimental): intra-alveolar placement of the hemostatic dressing ETIK COLLAGENE immediately after tooth extraction.
  Interventions: Device: Hemostatic dressing ETIK COLLAGENE
- Comparator (Other): the alveolus is left empty after tooth extraction.
  Interventions: Other: Comparator

INTERVENTIONS:
Device: Hemostatic dressing ETIK COLLAGENE — The hemostatic dressing ETIK COLLAGENE is placed in the alveolus immediately after tooth extraction. The presence of bleeding in the alveolus is assessed every 30 seconds for 8 minutes; then the surgical site is sutured.
  Arms: Device under investigation
Other: Comparator — The alveolus is left empty after tooth extraction. The presence of bleeding in the alveolus is assessed every 30 seconds for 8 minutes; then the dressing ETIK COLLAGENE is placed in the alveolus and the surgical site is sutured.
  Arms: Comparator

SUMMARY:
This study is a multicentric randomised (2 groups, ratio 1:1) Post Market Clinical Follow-up trial. 38 subjects (teeth) requiring a simple tooth extraction or multiple tooth extraction on the same quadrant and taking curative or preventive antithrombotic treatment will be included (19 in each group).

The aim of the study is to assess the efficacy of ETIK COLLAGENE (Topical hemostatic collagen-product) on the hemostasis (time to stop bleeding) after tooth extraction.

The hemostasis is measured by assessing the presence of bleeding within the first 8 minutes post-extraction.

Group 1: intra-alveolar placement of ETIK COLLAGENE immediately after tooth extraction.

Group 2: the alveolus is left empty after tooth extraction (the use of ETIK COLLAGENE is delayed 8 minutes after tooth extraction, before suture).

Subjects will be followed-up to 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age > 18 years old,
* Patient undergoing a simple tooth extraction or multiple tooth extraction on the same quadrant,
* Patient taking curative or preventive antithrombotic treatment or patient with a moderate thrombocytopenia,
* Patient reachable after surgery,
* Signed informed consent form,
* Subject affiliated to a health insurance system, or is a beneficiary.

Exclusion Criteria:

* Known allergy to bovine collagen,
* Preoperative INR<1.5 or >3 or instable,
* Patient with high risk of bleeding, history of postoperative hemorrhagic complication,
* Treatment with bone resorption inhibitor, or patient irradiated at the cervico-facial level,
* Contraindication to anesthesia using articaine with 1:200,000 epinephrine,
* Clinical follow-up expected to be difficult,
* Presence of uncontrolled hypertension, uncompensated diabetes or other clinically relevant systemic alterations,
* Current participation in another clinical trial or subject still within the exclusion period of a previous clinical trial,
* Vulnerable subjects.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2022-01-25 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2022-05-20 (Actual)

PRIMARY OUTCOMES:
Assessment of time to hemostasis after tooth extraction | over 8 minutes after tooth extraction
  For each patient, the time to stop bleeding (expressed in minutes) is assessed as follows : every 30 seconds from the tooth extraction (T0) to 8 minutes post extraction, the oral surgeon observes the alveolus during 5 seconds and records the presence or absence of bleeding.

SECONDARY OUTCOMES:
Rate of bleeding at 20 minutes | 20 minutes after tooth extraction
  % patients with bleeding occurring after suture, during the 10-minutes local compression period.
Occurrence of secondary post-extraction bleeding | 7 days
  Number of post-extraction bleeding
Level of pain after dental extraction by a numeric scale | At the end of the oral surgery, day 1, day 2, day 3
  The pain is assessed by patients in a diary using a numeric scale (range from 0 (= no pain) to 10 (= the worst pain)) each day from the end of the oral surgery to Day 3.
Number of adverse and serious adverse events | From the end of the oral surgery to Day 7
  Adverse events recorded from the tooth extraction to the end of follow-up visit will be used to assess the safety of hemostatic dressing and surgical procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Flora THIBAUT, DDS, Principal Investigator — Centre de soins dentaire CHU Rennes
Locations (2):
- France (2):
  - Faculté d'odontologie du CHU Nantes, Nantes
  - CSD Rennes, Rennes

IPD SHARING:
Plan to Share IPD: No